CLINICAL TRIAL: NCT02755701
Title: The Effect of Branched-chain Amino Acid on the Improvement of Serum Albumin Level in Cirrhotic Patients With Ascites: A Multi-center, Randomized, Double-blind, Placebo-controlled, Investigator Initiated Clinical Trial
Brief Title: The Effect of Branched-chain Amino Acid on the Improvement of Serum Albumin Level in Cirrhotic Patients With Ascites
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Collaborators: Severance Hospital (Other); Kyunghee University (Other); Wonju Severance Christian Hospital (Other); Korea University Anam Hospital (Other); Hanyang University (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Sang Gyune Kim, Associate professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIV_ACT Trial_I
Record Dates: First submitted 2016-04-21; First posted 2016-04-29 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Cirrhosis; Ascites
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCAA group (Experimental): Branched-chain amino acid, 4.15g, Tid
  Interventions: Drug: Branched-chain Amino Acid
- Placebo group (Placebo Comparator): Placebo, 4.15g, Tid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Branched-chain Amino Acid — BCAA (livact) will be administered 3 times a day during 24 weeks
  Other Names: Livact®
  Arms: BCAA group
Drug: Placebo — Placebo will be administered in the same way
  Arms: Placebo group

SUMMARY:
To compare the efficacy of branched-chain amino acid in serum albumin level in cirrhotic patients with ascites.

DETAILED DESCRIPTION:
Branched-chain amino acid (BCAA) is known to reduce the relapse rate of liver cancer as it is associated with insulin resistance and has been reported to improve the progression of liver fibrosis when used in combination with an angiotensin-converting enzyme. With regard to the effect of liver function improvement, in a research conducted in South Korea, approximately 41.2% of the patients showed recovery of the normal albumin level when BCAA was administered to them for about 10 weeks during radiation therapy for liver cancer. Additionally, in other overseas researches, the changes in the values of total protein and albumin were significantly smaller in the patients who underwent transarterial chemoembolization (TACE) to whom BCAA was administered than in those to whom BCAA was not administered.

The hypothesis of this study is that the serum albumin value will be increased significantly in the cirrhotic patients with ascites to whom BCAA is administered than the patients to whom placebo is administered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 and ≤ 70 years;
* Presence of liver cirrhosis
* Serum albumin level ≤ 3.5g/dl, ultrasound or CT scan confirmed ascites (≥Grade 1)
* No administration of diuretics and BCAA within the past 1 week
* Voluntary consent to take part in this trial

Exclusion Criteria:

* Child-Pugh score > 12
* Having been diagnosed as HCC within the past 5 years
* Serum creatinine > 1.5mg/dl
* Serum bilirubin > 5.0mg/dl
* Presence of such complications as SBP, or hepatic encephalopathy(West Haven grade ≥ 3)
* Patients who experienced organ failure by acute exacerbation of liver cirrhosis within the past 1 month
* Presence of serious cardiac or respiratory disease
* Contraindicated to either diuretics or BCAA
* Having commenced anti-viral treatment against hepatitis C, B within the past 1 month
* Pregnant or lactating women
* Chronic alcohol taker
* Woman patients who do not agree to the contraception from baseline to 12 month
* Unsuitable patients judged by investigator
* Patients participating in another clinical trial within 1 month

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum albumin level | 24 week

SECONDARY OUTCOMES:
Change in serum albumin level | 12 week
Rates of albumin normalization | 12, 24 week
Change in dose of diuretics | 12, 24 week
Improvement in terms of severity of ascites (International Ascites Club grade) | 24 week
Development rate of cirrhotic complications(including acute kidney injury, hepatic encephalopathy, variceal bleeding, peritonitis, etc) | 24 week
Improvement in Child-Pugh score, class | 24 week
Change in MELD, MELD-Na | 24 week
Improvement in sarcopenia | 24 week
Change in muscle mass | 24 week
Change in muscle strength | 24 week
Improvement in SF-36(short form-36) | 24 week
Change in HOMA-IR(homeostatic model assessment-insulin resistance) | 24 week

OTHER OUTCOMES:
Change in serum cystatin c | 12, 24 week
Change in HVPG(hepatic venous pressure gradient) | 24 week
Radiological characteristics of patients who have reaction to the branched-chain amino acid agent | 24 week
Change in serum creatinine | 12, 24 week
Improvement on PHES (psychometric hepatic encephalopathy score) | 24 week
Improvement on relative adrenal insufficiency | 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Sang Gyune Kim, Principal Investigator — Soon Chun Hyang University
Locations (8):
- Stanford University School of Medicine, Palo Alto, California, United States
- South Korea (7):
  - Wonju severance christian hospital, Wŏnju, Gangwon-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Kyunghee university hospital, Seoul
  - Korea university anam hospital, Seoul
  - Severance hospital, Seoul
  - Soonchunhyang university seoul hospital, Seoul
  - Hanyang university hospital, Seoul

IPD SHARING:
Plan to Share IPD: No